CLINICAL TRIAL: NCT06871319
Title: EVALUATION of the DIFFICULTY LEVELS of RESTORATIVE PROCEDURES of ENDODONTIC TREATED TEETH
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Sakine Sena Konstantoulas, Research Asistant, TC Erciyes University
Other Study IDs: EU-DHF-SSK-01
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Teeth with Root Canal Treatment
Keywords: restorations; root canal treatment
MeSH Terms: interventions — Radiography, Panoramic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: periapical x-ray, orthopantomography — Radiographic exams such as periapical x-rays and orthopantomography are necessary to evaluate the root canal system of teeth.

SUMMARY:
The goal of this observational study is to evaluate the difficulty levels of restorations of endodontically treated teeth. The main question it aims to answer is:

• Does the 8 predetermined criteria effect the difficulty levels of restorations of endodontically treated teeth.

Participants who has endodontically treated teeth or teeth to be treated endodontically, will undergo clinical and radiological examination. After that clinician will score the teeth between 1-6 based on predetermined criteria.

ELIGIBILITY:
Inclusion Criteria:

Patients who have at least one tooth with root canal treatment

Exclusion Criteria:

Patients who does not have any teeth with root canal treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who applied to Erciyes University Faculty of Dentistry, Department of Restorative Dentistry
Sampling Method: Probability Sample
Enrollment: 654 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
How hard is it to restore a tooth with root canal treatment based on 8 predetermined criteria. | At the time of enrollment
  For each criteria there are 6 scores. 1-2 are easy scores. 3-4 are medium scores. 5-6 are hard scores. This scores are decided by the clinician.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Melikgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No